CLINICAL TRIAL: NCT03924037
Title: Integrating Intergenerational Cultural Knowledge Exchange With Zero Suicide
Brief Title: Zero Suicide Plus KICKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Brandi C. Fink, PhD, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-031
Record Dates: First submitted 2019-04-15; First posted 2019-04-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Suicide; Suicidal Ideation; Suicidal Intention; Suicidal and Self-injurious Behavior
MeSH Terms: conditions — Suicide; Suicidal Ideation; Self-Injurious Behavior | interventions — Self-Help Groups

STUDY DESIGN:
Intervention Model Description: This study will utilize a between-subjects design with random assignment to the control (ZS) and the experimental groups (ZS+).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero Suicide (Active Comparator): Participants randomly assigned to the Zero Suicide arm will also participate in a weekly support group until the final follow-up time point when they will be crossed-over into the intergenerational knowledge sharing group.
  Interventions: Behavioral: Support group
- Zero Suicide plus KICKS (Experimental): Participants randomly assigned to the Zero Suicide plus KICKS arm will participate in a weekly intergenerational knowledge sharing group.
  Interventions: Behavioral: Intergenerational Knowledge Sharing group

INTERVENTIONS:
Behavioral: Intergenerational Knowledge Sharing group — Participants will attend a CBPR developed 12-session individual treatment for suicidal behavior. In addition to receiving the 12-session individual treatment, participants that are assigned to the Intergenerational Knowledge Sharing group will attend 12 weekly groups taught by tribal elders that focuses on sharing knowledge about the tribe.
  Arms: Zero Suicide plus KICKS
Behavioral: Support group — Participants will attend a CBPR developed 12-session individual treatment for suicidal behavior. In addition to receiving the 12-session individual treatment, participants that are assigned to the support group will attend 12 weekly support groups led by a behavioral health specialist that focuses on social support of the youth.
  Arms: Zero Suicide

SUMMARY:
Integrating Intergenerational Cultural Knowledge Exchange with Zero Suicide is an innovative study in a Southwestern tribal nation that incorporates Zero Suicide into Indian Health Services (IHS) primary care settings. The goal of this study is to determine the effectiveness of Zero Suicide plus a cultural component (ZS+) (experimental group) compared to Zero Suicide (ZS) alone (control group) on suicidal ideation, behaviors, and resiliency in a randomized control trial of 138 AI youth ages 12-24 at two rural IHS clinics on the Pueblo of San Felipe. The long-term goal of this study is to determine which is more effective at reducing suicidal ideation and behaviors and increasing resiliency, ZS+ or ZS alone. Year 1 will focus on training providers on the Zero Suicide model and manualizing the Katishtya Intergenerational Culture Knowledge Seminars (KICKS) curriculum that was piloted and positively evaluated over the past three summers as a cultural module to improve the adoption and acceptability of Zero Suicide. Years 2-4 will focus on participant recruitment, assignment to experimental and control groups, and implementation. Year 5 will focus on data analysis and dissemination. Data will be collected from all experimental and control group participants at 4 time points: baseline, 12-weeks, 6-months and 9-months to explore the effects of the intervention over time. The central hypothesis is that ZS+ will be more effective then ZS alone. The investigators propose three aims: (1) Specific Aim 1: Using Community Based Participatory Research (CBPR), partner with tribal stakeholders and researchers to formally manualize the KICKS cultural module for Zero Suicide (ZS+); (2) Specific Aim 2: To determine if adding a cultural component to the Zero Suicide model is more effective at reducing risk factors and increasing resiliency in AI youth than Zero Suicide alone; and (3) Specific Aim 3: Determine the essential features of the KICKS module for adaptation by other tribes and disseminate the model.

DETAILED DESCRIPTION:
Across the nation, suicide is the second leading cause of death in youth 10-24 years old. This public health crisis is particularly acute in American Indian (AI) communities where the suicide rate is 50% higher than that of non-Hispanic Whites. From 2009-2012, the age-adjusted suicide rate for American Indian/Alaska Native youth ages 10-24 years old was alarmingly higher than the overall rate for youth in this same age group nationally (14.66/100,000 vs. 8.25/100,000). In New Mexico (NM), the youth suicide rate is consistently at least 1.5 times the U.S. rate at 14.2/100,000, which is 75% higher than the national average. Importantly, NM has the highest proportionate AI population in the continental USA, and among the 22 tribes in NM the youth suicide rate is even greater (21.4/100,000). Also in NM, the percent of deaths due to suicide among AI youth by age range compared to all races is 29% vs.13% for ages 10-14, 32% vs.18% for ages 15-19, and 25% vs.16.5% for ages 20-24.3 The Pueblo of San Felipe, a tribal nation in NM and the target population for the proposed study, has incredibly high rates of suicidal ideation and behavior with 21.8% of students reporting that they seriously considered suicide, 14.9% reporting that they made a suicide plan, and 11.6% reporting that they attempted suicide in the past year compared to 19%, 11.3%, and 7% respectively statewide. A recent school needs assessment of over 300 students found even higher rates, as 40% of youth expressed feeling frequently depressed within the last year, 17% reported feeling sad or depressed most or all of the time within the last month, and 30% noted they attempted suicide one or more times within the last month. Thus, suicide is of grave concern to tribal communities in NM, especially the Pueblo of San Felipe, and developing systematic strategies for reducing suicide among AI youth is of utmost importance.

Risk Factors Associated with Youth Suicide. The probability of attempting suicide has been found to dramatically increase as the number of risk factors increases. Research on suicidal behavior in youth indicates that the odds of experiencing suicidal ideation and/or suicide attempts are nearly three times more likely if the youth is using alcohol. Even more concerning is that the odds of a completed suicide are five to 13 times greater for youth diagnosed with a substance use disorder.6 Furthermore, lethality of suicide attempts increases with alcohol use, and 40% of suicide attempts and 37% of suicides preceded by acute use of alcohol. While depression is associated with suicidal behavior, depression predicts suicide attempts significantly less well when controlling for substance use. Similarly, exposure to violence, including domestic and intimate partner violence, increases the probability of suicidal ideation and behaviors, as does historical trauma (defined as the cumulative emotional and psychological wounding across generations which emanates from massive group trauma). Unfortunately, AI youth experience exceptionally high rates of these risk factors, including substance abuse, exposure to violence, and the profound repercussions of historical trauma (domestic violence, abuse, etc.). The proposed study addresses risk factors by incorporating these topics into the cultural component of the intervention known as Katishtya Intergenerational Culture Knowledge Seminars (KICKS), as they are NOT addressed in Zero Suicide.

Resiliency as a Buffer. Resilience is also a critical component of suicide prevention. Buffering is the idea that having resources, such as social support or cultural grounding, can mitigate against adverse stressful events.16 The Buffering Hypothesis is a model linking resilience to suicidality that focuses on beliefs, which buffer individuals in the face of stressors. Resilience factors are viewed as existing on a separate dimension to risk which act to moderate the impact of suicidality. The presence of these factors results in resilience and the absence increases risk for suicidality. Resiliency factors include internal protective factors (positive beliefs or feelings about oneself and satisfaction with life), external protective factors (ability to seek resources helpful when faced with personal difficulties), and emotional stability (positive beliefs about one's ability to regulate suicide-related thoughts and behaviors when confronting emotionally distressing events). Importantly, research shows that increasing protective factors can be more effective at reducing the probability of suicide attempts for AI youth then decreasing risk factors, and other studies indicate that interventions are only effective to the extent that they recognize and promote AI cultural values, traditional practices, and cultural identity development. Thus, to improve suicide prevention program acceptability and adoption it is critical to include culturally relevant strength-based and resilience focused components to suicide prevention models.

Relationship between Suicide and Health Disparities. Health disparities are "preventable differences in the burden of disease, injury, violence, or opportunities to achieve optimal health that are experienced by socially disadvantaged populations". Barriers to mental health care utilization for AI youth include: lack of culturally competent treatment providers, a general mistrust in services provided within a Western medical model, and personal experiences of discrimination in health care settings. These barriers have been found to reduce the likelihood of seeking care, even when suicidal ideation or behaviors are present, thus, contributing to the higher incidence of youth suicide in AI communities. The proposed study addresses disparities in access and acceptability by adding a cultural component to the Zero Suicide model.

Call to Develop and Test Innovative Suicide Prevention Models. In 2014, the National Action Alliance for Suicide Prevention's Research Prioritization Task Force published strong recommendations regarding the need to develop and test feasible and effective suicide prevention interventions. Although there have been considerable studies focusing on youth suicide prevention there is insufficient evidence to know which strategies are most effective in preventing suicide among AI populations. Importantly, AI adolescents experience significant risk factors for suicide, including substance abuse and exposure to violence (e.g., physical and sexual violence, domestic violence, intimate partner violence, and premature death of relatives due to violence, accidents, or suicide).5 Although suicide prevention has been shown effective in reducing suicidal ideation and behaviors with youth, there are limited Randomized Control Trials (RCTs) focused on preventing suicide attempts in AI youth populations, thus it is unclear whether the results of previous studies are generalizable. Critically, examining the effect of suicide prevention interventions in AI primary care settings is vital as the majority of individuals who die by suicide (80%) have contact with a primary care clinician or Emergency Department (ED) in the year prior to death. There is promising research on the effectiveness of Zero Suicide (ZS), a population-based model implemented through a large HMO system in the Midwest. However, ZS has not been studied with AI populations or in tribally-based Indian Health Service (IHS) primary care settings. Additionally, ZS does not include culturally-adapted interventions, which have been found to produce larger effect sizes than un-adapted interventions for minority populations.

The Zero Suicide Model. ZS is a population health-based approach to suicide prevention underscoring the belief that suicide deaths are preventable and that individuals are often not recognized in fragmented, busy health care systems.27 Studies of the Perfect Depression Care program, the precursor to ZS, showed significant findings including an 82% decrease in suicide deaths between baseline and intervention in a large urban Midwest health System. ZS has seven essential elements for health care systems, including: (1) Lead- create a leadership-driven, safety-oriented culture committed to reducing suicide for people under care; (2) Train- develop a workforce that understands and responds to depression and suicidal behaviors; (3) Identify- universally screen and assess suicide risk; (4) Engage- ensure every individual has timely and adequate pathways to care and includes a brief safety plan (5) Treat- use effective, evidence-based treatment, such as Cognitive Behavioral Therapy-Suicide Prevention (CBT-SP), to target suicidal ideation and behaviors; (6) Transition- provide continuous contact and support, especially after acute care; and (7) Improve- apply a data-driven quality improvement approach to inform system change and improve patient outcomes. The ZS toolkit provides resources on these elements, including training manuals, an organizational self-study, work plan template, and consumer engagement strategies. The need for consideration of cultural adaptation is indicated (zerosuicide.sprc.org) but not specified.

Importantly, data is available on the effectiveness of each of the ZS elements. For instance, training with booster sessions for healthcare professionals in primary care and ED settings has been found to improve identification of suicide warning signs and willingness to refer patients for mental health services, and to reduce suicidal behavior in situations where the roles of gatekeepers are formalized and access to treatment is readily available. Findings also support the importance of integrating brief universal screening in primary care settings to quickly identify at-risk individuals and prompt healthcare professionals to make referrals. Research found that there was a four-fold increase in the detection of suicidal ideation by pediatricians when screening tools were used in outpatient clinics. Additionally, pediatric ED studies show screening for suicide risk can reveal previously undetected suicidal ideation in youth presenting with medical complaints. Importantly, screening must confidently rule out patients with no appreciable risk, and balance feasibility with effectiveness. Finally, research supports the importance of feasible and acceptable treatment such as CBT-SP for those identified as being at risk for suicidal ideation or behaviors. CBT-SP has been found to result in a greater reduction of suicidal ideation than treatment as usual, and consists of a chain analysis of the index suicide attempt, and development of a safety plan and individualized treatment plan to reduce reattempts.

Implementation of ZS in AI Communities is NOT Enough. Importantly, implementing ZS in tribal communities requires cultural adaptation. As noted earlier, culturally-adapted interventions have been found to produce larger effect sizes than un-adapted interventions for minority populations. In addition, research indicates that substance abuse and exposure to trauma are significant risk factors impacting suicide in AI youth. Finally, strengthening protective factors may be more important than reducing risk factors in addressing suicide for AI youth. ZS does not focus on reducing risk factors and increasing resiliency. The proposed study incorporates all of these elements into the KICKS component, thereby increasing the appropriateness and acceptability of ZS for AI populations.

Importance of Cultural Adaptations to Improve Suicide Outcomes among AI Youth. For ZS to be adopted, implemented, and sustained in tribal communities, cultural consideration is critical. Two large studies found that for AI youth strengthening protective factors may be more important than reducing risk factors in addressing suicide, and mentoring from parents, extended family, teachers, and friends helps AI youth overcome failure, succeed in school, and develop resiliency. Engaging youth in teachings on traditional narratives, beliefs and practices, and intergenerational approaches that focus on communication and awareness across generations have also been found to increase resiliency. Moreover, research demonstrates that elders play a critical role in fostering resilience by providing mentoring, teaching, and social support to AI youth through transmission of valuable cultural beliefs, traditions, and practices. The proposed study incorporates all of these elements to reduce suicidal ideation and behaviors and increase resiliency.

Katishtya Intergenerational Culture Knowledge Seminars (KICKS) Cultural Adaptation. The cultural adaptation proposed in this study is the Katishtya Intergenerational Culture Knowledge Seminars (KICKS), an intergenerational program to promote resiliency and positive connections between San Felipe youth and elders. Over the past three years, San Felipe developed and piloted KICKS, where elders share traditional culture, language, lifeways, and history with San Felipe youth in an eight-week daily seminar. KICKS was developed to improve resiliency through exposure to intergenerational cultural teachings, and preliminary data indicates that over 90% of youth felt they acquired substantial knowledge of each of the traditional activities, indicating that KICKS fostered learning and resiliency. Well received by tribal members and tribal leadership, KICKS is a perfect cultural module to increase resiliency and improve acceptability and adoption of ZS.

Partnership as a Predictor of Behavioral Health Outcomes. Another potential variable is the quality of stakeholder partnerships. In the last decade, the literature on CBPR has moved beyond a focus on partnership processes and improved success at recruiting participants, to recognizing the significant evidence of its impact on health outcomes. Adherence to CBPR principles and strategies show positive impacts on health behavior, self-efficacies, perceived social support, empowerment, and improved health status; as well as improved policies to reduce health inequities. Mental health outcomes in particular have been shown in the community engagement arm of an extensive RCT. UNM's ten-year study on quantitative and qualitative methods to assess partnering processes and their associations with outcomes will prove invaluable for measuring the quality and impact of the community partnership in San Felipe. These assessments will be critical to determine the partnership's impact on the identified outcomes. They will also support a mutual iterative learning process that will contribute to ongoing research capacity building within the tribe itself for greater sustainability of the intervention over time.

Benefits of Transdisciplinary, Multi-Level and Multi-Domain Interventions. Finally, in perfect alignment with the mission of the Transdisciplinary Research, Equity and Engagement Center for Behavioral Health (TREE Center), Integrating Intergenerational Cultural Knowledge Exchange with Zero Suicide is a transdisciplinary, multi-level suicide prevention intervention study that addresses resiliency and risk factors related to AI youth suicidal ideation and behaviors. Effective health disparities interventions benefit from transdisciplinary, multi-level and multi-domain components. The transdisciplinary research team represents disciplines across the University (e.g., Psychology, Psychiatry, Public Health, Clinical and Translational Sciences) as well as community partners across child-serving tribal programs (e.g., Primary Care, Behavioral Health, Education, Social Services) collaborating on the creation of an innovative AI youth suicide prevention model. This also study employs a multi-level intervention approach. The first level is the Individual level (youth who receive universal screens and participate in the ZS or ZS+ intervention). The second is the Group level (KICKS is provided in a group format), and the third is the Community level (elders who participate in the KICKS module, school impacted by providing universal screens at the SBCH, and larger community impacted through ZS implementation in all primary care settings). This multi-level approach enables us to understand issues of inequities in health and monitor the outcome of the intervention across levels. This study also aims to reduce behavioral health disparities by simultaneously addressing the needs and stressors of AI youth across multiple domains including behavioral, sociocultural and health care system.

Summary. Because suicide is a low base rate behavior, very large samples are needed to conduct adequately powered suicide prevention trials. Suicidal ideation and behavior, however, are often warning signs of completed suicide, making it especially important to target in intervention studies. Given the research supporting ZS and the fact that Indian Health Services (IHS) identified "Zero Suicide [as] a call to relentlessly pursue a reduction in suicide for those who come to us for care," there is a clear recognition that ZS is a promising practice for tribal behavioral health. However, resilience-focused approaches, such as KICKS, must be included, as must reduction of risk factors related to substance abuse and violence. Thus, the current proposal will examine differences in reducing suicidal ideation and behaviors, and increasing resiliency for AI youth who participate in ZS vs. ZS+.

APPROACH Study Overview. The proposed project will manualize the KICKS module and then conduct a Randomized-Controlled Trial (RCT) of Zero Suicide (ZS) and Zero Suicide plus Katishtya Intergenerational Culture Knowledge Seminars (ZS+) in AI youth ages 12-24 years old from the Pueblo of San Felipe. It is transdisciplinary and multi-level collaborative research project between the University of New Mexico, the Pueblo of San Felipe, IHS clinics; and community stakeholders (e.g., youth, elders, family members, health care providers, tribal leadership).

Community Advisory Committee. The investigators will form a Community Advisory Committee (CAC) for this study in San Felipe comprised of tribal program representatives from Behavioral Health, Primary Care, Social Services, Schools, Recreation, Tribal Leadership, UNM researchers, other stakeholders. Dr. Altschul (MPI) and Ms. Tenorio (PD) will use a CBPR approach to co-facilitate the CAC and guide all aspects of the study including, refining data collection methods, participant recruitment, implementation, data analysis, and dissemination. One CAC member will also serve on the NM TREE Center Community Scientific Advisory Council.

Specific Aim 1: Using CBPR, partner with tribal stakeholders and researchers to formally manualize the KICKS cultural module for Zero Suicide (ZS+). The objective of Specific Aim 1 is to develop a manual for the KICKS cultural module of ZS+ using a CBPR approach. To obtain this objective the investigators will develop a community-based workgroup, the KICKS Review Committee, to collaboratively formalize the KICKS module. The rationale for this Aim is that having a manualized intervention will increase fidelity to the KICKS module, and ensure delivery that is culturally appropriate, feasible, and effective. When the proposed research for this Aim has been completed, the investigators expect to have a formalized manual that will be used to consistently implement KICKS and to test Specific Aim 2 to compare implementation of ZS+ vs. ZS alone in the San Felipe IHS clinics.

Research Design and Method. KICKS was developed in 2014 for youth to see that cultural knowledge is key to resiliency, language is vital to maintain traditions, and Native people were given many gifts from the Creator, including natural supports and protective factors, that enabled their survival for centuries. Youth and elders met daily for 8-weeks and participated in Keres language instruction, traditional storytelling, Pueblo history, traditional dances, crafts, and visiting traditional and cultural sites. Youth learned about proper introductions using AI name and clan; the traditional naming process; family extensions/kinship; types and uses of corn; Pueblo history including emergence, migration and settlement; traditional prayer; clan responsibilities; traditional crafts (pouches, arrows, dance regalia); language and item identification; respect, acknowledgement, acts of kindness, and cultural responsibilities; traditional dances, including regalia identification/significance; and traditional cooking, sewing, and pottery making. In exchange, youth taught elders about modern technology, including email access, use of iPads, etc. This intergenerational knowledge sharing created positive outcomes for both youth and elders, including increased self-reported resiliency.

Development of the KICKS module will occur through the KICKS Review Committee, including the KICKS Coordinator, elders and youth who participated in the KICKS pilot, university researchers, and other interested parties. The Committee will meet twice monthly for 8 months to review agendas from the KICKS pilot, discuss successes and challenges noted during the pilot, identify core content areas, consider potential additions, and discuss flow of the curriculum. Although there are agendas for each KICKS session, it is important to manualize the program so that the module can be followed with fidelity throughout the study. In addition, certain topics, such as historical trauma and substance abuse, were not explicitly included but will be added due to their importance as potential risk factors for suicidality. This process will use CBPR strategies to ensure collaboration with community partners during all phases of research, including study design, implementation, data collection, interpretation, and dissemination. UNM data collectors will gather detailed qualitative meeting minutes to document progress made and identify themes that emerge for inclusion in the manual. The final manual will be presented to Tribal Leadership and the Tribal Council for review and approval. This CBPR process recognizes the significance of culture in research design and implementation to facilitate relevance to the community, ethical conduct, external validity, and effectiveness.

Specific Aim 2: To determine if adding a cultural component to the Zero Suicide model (ZS+) is more effective at reducing risk factors and increasing resiliency in AI youth than Zero Suicide alone (ZS). The objective of Specific Aim 2 is to assess the effectiveness of ZS enhanced with a cultural module (ZS+) compared to ZS alone at reducing suicidal ideation and behaviors and increasing resiliency. To achieve this objective, the investigators will test the working hypothesis that ZS+ will be more effective then ZS alone in reducing suicidal ideation, behaviors and attempts. The rationale for Aim 2 is that successful completion of the proposed research will contribute a missing, fundamental element to the suicide prevention knowledge base critical to the development of a youth suicide prevention program designed and tested with AI youth and found to be culturally appropriate, feasible, and effective. Achieving these outcomes will collectively inform the suicide prevention field about the effectiveness and feasibility of implementing ZS and ZS+ in IHS primary care settings, and provide a greater understanding of the potential mechanisms that reduce suicidal ideation and behaviors and increase resiliency for AI youth, a much-needed finding in Indian Country. Achieving these outcomes will also inform the field about the adoption and acceptability of the ZS model; and whether the quality of the community stakeholder partnership is a predictor of behavioral health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* American Indian youth aged 13-24 years old who are San Felipe tribal members living in the Pueblo
* Endorse suicidal ideation or behaviors on a universal screen by their primary care provider.

Exclusion Criteria:

* Younger than age of 13 years old or
* Older than the age of 24,
* Not American Indian,
* Youth who do not receive health services at either of the IHS clinics at the Pueblo of San Felipe,
* Youth who screen negative for suicidal ideation and/or behavior,
* Refuse to participate in the study, and/or
* Cognitively unable to provide informed consent as demonstrated by a brief cognitive screen prior to completion of the baseline interview.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 222 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction in suicidal behavior | 12 weeks
  The individual treatment sessions will result result in a change in suicidal behavior as measured by the Suicidal Behaviors Questionnaire - Revised and the Suicide Ideation Questionnaire at baseline to the completion of individual treatment sessions.
Improvement in resilience | 12 weeks
  The Intergenerational Knowledge Sharing group should result in a change in youth resilience as measured by the Suicide Resilience Inventory-25 at baseline to the completion of the KICKS group sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Altschul, PhD, Principal Investigator — University of New Mexico; Brandi C Fink, PhD, Principal Investigator — Oklahoma University Health Sciences Center
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States